CLINICAL TRIAL: NCT04466202
Title: The Effect of Music With Structured Verbal Training on Pain, Anxiety and Satisfaction During Prostate Biopsy
Brief Title: Effectiveness of the Music With Structured Verbal Training During Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, RN, PhD, Asst Prof, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020.02.13-07
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Pain; Anxiety; Satisfaction; Urological Nursing
Keywords: Anxiety; Nursing; Pain; Satisfaction; Prostate biopsy
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group with Structured Verbal Training (Experimental): Music with structured verbal training was applied during transrectal ultrasound guided prostate biopsy.
  Interventions: Other: Music with Structured Verbal Training
- Control Group (No Intervention): The control group did not listen to music during the procedure, and they received routine training.

INTERVENTIONS:
Other: Music with Structured Verbal Training — Structured verbal training on prostate biopsy was given to the intervention group before the procedure, and then patients in this group listened to the music they preferred during the procedure with headphones.
  Arms: Music Group with Structured Verbal Training

SUMMARY:
Transrectal ultrasound (TRUS) guided prostate biopsy is a gold standard method widely used in the diagnosis of prostate cancer. This procedure can be very painful and anxious for men. Various pharmacological methods can be used to relieve patients' pain and discomfort during TRUS-guided prostate biopsy. Although there is still no consensus on the solution suggestions for pain and anxiety due to biopsy, it is known that music, which is a non-pharmacological method, is effective in this regard. The aim of this study is to evaluate the effect of music with structured verbal training on patients' pain, anxiety and satisfaction levels during transrectal ultrasound-guided prostate biopsy.

DETAILED DESCRIPTION:
Although there have been several studies examining the effect of music on pain and / or anxiety during TRUS prostate biopsy, only one study has been found examining the effect of stress management (music and one-to-one simulation training) on patients' pain and anxiety levels. In addition, there is only one study on the effectiveness of the training method (written and video-based training) on anxiety levels of patients related to prostate biopsy. For this reason, it is thought that music will be more effective on pain and anxiety levels along with structured verbal training to alleviate the discomfort associated with patients' biopsy procedure.

ELIGIBILITY:
Inclusion Criteria:

* being over the age of 40
* male gender
* transrectal ultrasound guided prostate biopsy for the first time
* agreeing to participate in the study

Exclusion Criteria:

* presence of any contraindication for prostate biopsy
* any analgesic used 24 hours before prostate biopsy

Ages: 40 Years to 86 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
change on pain intensity as measured by Visual Analog Scale | "just before procedure", "during procedure" and "5 minutes after procedure"
  The average score change on pain intensity as measured by Visual Analog Scale. This scale is an unidimensional measure commonly used to measure pain intensity. The scale is a measuring tool with length of 0-10 cm (0-100 mm). High scores on the scale indicate that pain intensity is high.

SECONDARY OUTCOMES:
score change on anxiety level as measured by State-Trait Anxiety Inventory | "just before procedure" and "5 minutes after procedure"
  The average score change on anxiety level as measured by State-Trait Anxiety Inventory. This scale is used to measure anxiety. The scores on the scale ranges from 20 to 80. The high scores on the scale indicate that anxiety is high.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Chang YH, Oh TH, Lee JW, Park SC, Seo IY, Jeong HJ, Kwon WA. Listening to music during transrectal ultrasound-guided prostate biopsy decreases anxiety, pain and dissatisfaction in patients: a pilot randomized controlled trial. Urol Int. 2015;94(3):337-41. doi: 10.1159/000368420. Epub 2014 Dec 18. PMID 25531837
- [Background] Chiu LP, Tung HH, Lin KC, Lai YW, Chiu YC, Chen SS, Chiu AW. Effectiveness of stress management in patients undergoing transrectal ultrasound-guided biopsy of the prostate. Patient Prefer Adherence. 2016 Feb 11;10:147-52. doi: 10.2147/PPA.S96991. eCollection 2016. PMID 26929606
- [Background] Cho SW, Choi HJ. Effect of Music on Reducing Anxiety for Patients Undergoing Transrectal Ultrasound-Guided Prostate Biopsies: Randomized Prospective Trial. Urol J. 2016 Apr 16;13(2):2612-4. PMID 27085561
- [Background] Chopra S, Rowe EW, Laniado M, Patel A. A prospective study analysing the effect of pain on probe insertion, and the biopsy strategy, on the patients' perception of pain during TRUS-guided biopsy of the prostate. N Z Med J. 2008 Dec 12;121(1287):39-43. PMID 19098966
- [Background] Packiam VT, Nottingham CU, Cohen AJ, Eggener SE, Gerber GS. No Effect of Music on Anxiety and Pain During Transrectal Prostate Biopsies: A Randomized Trial. Urology. 2018 Jul;117:31-35. doi: 10.1016/j.urology.2018.04.014. Epub 2018 Apr 27. PMID 29709434
- [Background] Tsivian M, Qi P, Kimura M, Chen VH, Chen SH, Gan TJ, Polascik TJ. The effect of noise-cancelling headphones or music on pain perception and anxiety in men undergoing transrectal prostate biopsy. Urology. 2012 Jan;79(1):32-6. doi: 10.1016/j.urology.2011.09.037. PMID 22202544